CLINICAL TRIAL: NCT05207644
Title: Letrozole and Misoprostol for Termination of Pregnancy up to 63 Days' Gestation: A Pilot Study to Evaluate the Safety and Acceptably of a User-friendly Regimen
Brief Title: Letrozole and Misoprostol for Termination of Pregnancy up to 63 Days' Gestation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1048
Record Dates: First submitted 2021-12-09; First posted 2022-01-26 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Pregnancy
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Letrozole followed by misoprostol (Other): There is only one arm in this study.
  Interventions: Drug: 30 mg letrozole followed by 800 mcg misoprostol

INTERVENTIONS:
Drug: 30 mg letrozole followed by 800 mcg misoprostol — 30 mg letrozole on day 1 followed by 800 mcg misoprostol on day 3

SUMMARY:
Study to determine if a user-friendly medical abortion regimen using letrozole and misoprostol is safe and acceptable.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy ≤ 63 days gestational age by ultrasound seeking termination of pregnancy
* Pregnancy visible on ultrasound
* Speaks English or Spanish
* Willing and able to return for follow-up appointment

Exclusion Criteria:

* People with gestations > 63 days gestational age
* Confirmed or suspected ectopic pregnancy or undiagnosed adnexal mass
* Pregnancy of unknown location
* IUD or contraceptive implant in place
* History of allergy to letrozole or misoprostol
* Unable to return for clinic-based follow-up
* Currently breastfeeding
* Twin or multiple pregnancy
* History of liver disease or abnormal liver function

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Safety Profile of medical abortion regimen | 2 weeks
  To evaluate the safety profile of a user-friendly letrozole-misoprostol regimen.

CONTACTS AND LOCATIONS:
Overall Officials: Tara Shochet, PhD, MPH, Principal Investigator — Gynuity Health Projects; Beverly Winikoff, MD, MPH, Principal Investigator — Gynuity Health Projects; David Turok, MD, MPH, Principal Investigator — The University of Utah
Locations (1):
- Planned Parenthood Salt Lake Health Center, Salt Lake City, Utah, United States